CLINICAL TRIAL: NCT04058899
Title: Dexmedetomidine Versus Nalbuphine in Prevention of Emergence Agitation Following Adenotonsillectomy in Pediatrics
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Elsayed Elagamy, Assisstant proffesor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Use of dexmedetomidine
Record Dates: First submitted 2019-07-29; First posted 2019-08-16 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Emergence Delirium
Keywords: dexmedetomidine; emergence agitation; adenotonsillectomy
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Nalbuphine; Infusion Pumps

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 groups ,dexmedetomidine group (DEX)group who will receive 0.5 µg/kg dexmedetomidine diluted in 50 ml of normal saline 0.9% to be given by IV infusion over 10 minutes after induction of anesthesia then 5ml of 0.9% normal saline IV ,nalbuphine group (NAL)group will receive IV infusion of 50 ml of 0,9%normal saline by IV infusion over 10 minutes then 0.1mg/kg nalbuphine diluted in 5ml of 0.9%normal saline IV after induction of anesthesia.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- , Dexmedetomidine group(DEX group) (Active Comparator): dexmedetomidine group (DEX)group who will receive 0.5 µg/kg dexmedetomidine diluted in 50 ml of normal saline 0.9% to be given by IV infusion over 10 minutes after induction of anesthesa then 5ml of 0.9% normal saline IV ,
  Interventions: Drug: Dexmedetomidine; Device: infusion pump
- Nalbuphine group(NAL group) (Active Comparator): nalbuphine group (NAL)group will receive IV infusion of 50 ml of 0,9%normal saline by IV infusion over 10 minutes then 0.1mg/kg nalbuphine diluted in 5ml of 0.9%normal saline IV after induction of anesthesia.
  Interventions: Drug: Nalbuphine; Device: infusion pump

INTERVENTIONS:
Drug: Dexmedetomidine — sedative and might be analgesic drug
  Arms: , Dexmedetomidine group(DEX group)
Drug: Nalbuphine — agonist antagonist narcotic
  Arms: Nalbuphine group(NAL group)
Device: infusion pump — infusion pump for titration of fluid containing drug infusion

SUMMARY:
The aim of the present study is to compare the effect of IV infusion 0.5 µg/kg dexmedetomidine and IV 0.1 mg/kg nalbuphine in preschool children for prevention of emergence agitation after adenotonsillectomy under sevoflurane anesthesia.

DETAILED DESCRIPTION:
Consent will be obtained from legal guardian of children,patients will be randomized according to computer randomization to one of two groups, dexmedetomidine group (DEX)group who will receive 0.5 µg/kg dexmedetomidine diluted in 50 ml of normal saline 0.9% to be given by IV infusion over 10 minutes after induction of anesthesia then 5ml of 0.9% normal saline IV ,nalbuphine group (NAL)group will receive IV infusion of 50 ml of 0,9%normal saline by IV infusion over 10 minutes then 0.1mg/kg nalbuphine diluted in 5ml of 0.9%normal saline IV after induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children of (American Society of Anesthesiologist)ASA physical status grade I or II.
* Aged 2-5 years
* Undergoing elective adenotonsillectomy.

Exclusion Criteria:

* History of hypersensitivity to the studied drug.
* Refusal of the legal guardian to participate in the study.
* Severely agitated child at induction of anesthesia
* Occurrence of postoperative bleeding at(Post Anesthesia Care Unit) PACU

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
postoperative agitation prevention in pediatrics after adenotonsillectomy under sevoflurane anesthesia | stay in postoperative care unit till discharge of patient to ward.Time frame is up to 24 weeks
  during stay in postoperative care unit using pediatric anesthesia emergence delirium score (PAED) as score equal or more than 16/20 is considered presence of agitation. during stay in postanesthesia care unit,score will be documented every 10 minutes by recovery staff.

SECONDARY OUTCOMES:
sedation in early postopertive time during child stay in postanesthesia care unit | stay in postoperative care unit till discharge of patient to ward.Time frame is up to 24 weeks
  stay in postoperative care unit using Ramsay sedation score evey 10 minutes till discharge to ward,assessed by recovery staff..Presence of score 4/6 or more means that child is sedated,and needs more time in recovery,..

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt